CLINICAL TRIAL: NCT01753609
Title: Safety and Performance Evaluation of TrimWeight Device - an Intragastric Auto-inflating & Degradable Balloon in a Swallow-able Capsule ("the Device"), for Enhancing Satiety and Satiation in Healthy Over Weight and Obese Volunteers
Brief Title: Safety and Performance Evaluation of Tulip Device in Healthy Overweight and Obese Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tulip Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TULIP-PRT-002-05-B-CTIL
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Over Weight; Obesity
Keywords: Over weight; Obesity
MeSH Terms: conditions — Obesity | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tulip capsule (Experimental): swallowing Tulip capsule for up to 29 days
  Interventions: Device: Tulip capsule

INTERVENTIONS:
Device: Tulip capsule — swallowing Tulip capsule for up to 29 days

SUMMARY:
The study will assess the safety and performance of an intragastric auto-inflating and degradable balloon

DETAILED DESCRIPTION:
The study will assess the safety and performance of an intragastric auto-inflating and degradable balloon, packed in a swallow-able capsule, in healthy subjects with 30 < BMI≤ 35.

ELIGIBILITY:
Inclusion Criteria:

* 21 ≤ Age <65 years
* 30 < BMI ≤ 35 kg/m2
* Healthy without any medication;
* No history of weight reduction of more than 5% of total body weight in the past 6 months;
* Normal blood count and chemistry;
* Hemoglobin level over 11;
* At least 3 bowel movements per week;
* Subject declares that he/she is able to go through gastroscopic examination;
* Subject is able and willing to give informed consent and follow protocol procedures.

Exclusion Criteria:

* Any history or evidence of significant cardiac, renal, neurologic, metabolic, pulmonary, gastrointestinal, hematologic abnormality, chronic hepatic disease or any other disease which in the judgment of the investigator would interfere with the study or confound the results;
* History or evidence of any active liver disease. (abnormal liver functions: >1.5 times upper limit);
* History or symptoms of thyroid disease which is not controlled by medication;
* Abnormal gastrointestinal findings: Diaphragmatic hernia > 3 cm; Active peptic ulcer; Erosive gastritis; Gastric outlet obstruction;
* Subject with IBD
* Significant swallowing disorders;
* Past history of any gastrointestinal surgery (excluding uncomplicated appendectomy);
* Malabsorption disorders.
* Is taking medications that reduce gastric acidity
* Currently using pharmaceutical agents or food supplements for weight loss;
* History of or current eating disorder such as anorexia or bulimia or compulsory overeating.
* History of food Allergy;
* Subject with poor venous access;
* Is taking chronic aspirin or other non-steroidal anti-inflammatory agents, or other medications known to be gastric irritants;
* Have any coagulation problem and/or taking any anticoagulant medications;
* Evidence of current malignant disease;
* Have history of any acute disease (viral, bacterial, pain, accident) in the last 6 weeks.
* Female subject who are breastfeeding or have a positive pregnancy test at screening or at any time during the study;
* Inability to give written informed consent;
* History of alcohol or drug abuse within 6 months of screening;
* Mental disorders;
* Currently participating in an ongoing clinical study
* Any reasons making the patient a poor candidate in the opinion of the investigator.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-03 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with device related serious adverse events | 36 days
  Safety will be assessed descriptively by summarizing device related SAEs, gastroscopic examination, daily diary, vital sign measurements, physical examination and abdomen circumference.

SECONDARY OUTCOMES:
Patient assessment of capsule tolerability | 36 days
  Comfort and tolerability will be assessed by the patient and will be recorded in a daily diary. Tolerability evaluation will include: assessment of swallow ability, gastrointestinal comfort, defecation effort, appetite.
Satisfying evacuation of the balloon from the stomach after oral intake | 36 days
  Number of subjects showing satisfying evacuation of the balloon from the stomach after oral intake by means of a gastroscopic examination

CONTACTS AND LOCATIONS:
Overall Officials: Sigal Fishman, Dr., Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center , Gastroenterology - Institute, Tel Aviv, Israel